CLINICAL TRIAL: NCT02353039
Title: Double Blind, Multicenter, Randomized, Placebo-controlled, Parallel-group, Phase II Study to Evaluate the Efficacy and Safety of GC6101A in Subjects With Gastritis
Brief Title: Phase II Study to Evaluate the Efficacy and Safety of GC6101A in Subjects With Gastritis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Green Cross Corporation (Industry)
Collaborators: C&R Research, Inc. (Industry); CRScube (Unknown)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GC6101A_P2
Record Dates: First submitted 2015-01-27; First posted 2015-02-02 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Gastritis
MeSH Terms: conditions — Gastritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- GC6101A 37.5mg (Experimental): Administer 12.5mg of GC6101A t.i.d for 2 weeks.
  Interventions: Drug: GC6101A 37.5mg
- GC6101A 75mg (Experimental): Administer 25mg of GC6101A t.i.d for 2 weeks.
  Interventions: Drug: GC6101A 75mg
- GC6101A 150mg (Experimental): Administer 50mg of GC6101A t.i.d for 2 weeks.
  Interventions: Drug: GC6101A 150mg
- Placebo (Placebo Comparator): Administer placebo t.i.d for 2 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GC6101A 37.5mg — Administer 12.5mg of GC6101A t.i.d for 2 weeks.
  Arms: GC6101A 37.5mg
Drug: GC6101A 75mg — Administer 25mg of GC6101A t.i.d for 2 weeks.
  Arms: GC6101A 75mg
Drug: GC6101A 150mg — Administer 50mg of GC6101A t.i.d for 2 weeks.
  Arms: GC6101A 150mg
Drug: Placebo — Administer placebo t.i.d for 2 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the investigational products in the patients with gastritis during their participation in the study.

DETAILED DESCRIPTION:
GC6101A is botanical drug products made from the Lonicerae Flos. Two hundred volunteers will participate in the study, receive 2-week treatment with GC6101A or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age is over 19 years old, men or women
* Patients diagnosed with acute or chronic gastritis by gastroscopy
* Patients with one or more erosions found by gastroscopy
* Signed the informed consent forms

Exclusion Criteria:

* Patients who is impossible to receive gastroscopy
* Patients with peptic ulcer and gastroesophageal reflux disease
* Patients with gastroesophageal surgery and surgery to reduce the secretion of gastric acid (Except for surgery for perforated peptic ulcer and cecectomy)
* Patients with esophageal varix
* Patients with malignant neoplasm of gastrointestinal tract
* Patients with thrombosis or administered with anti-thrombotic drugs
* Patients with consumption coagulopathy
* Patients administered with H2 receptor antagonists, muscarinic receptor antagonists, gastrin receptor antagonist, proton pump inhibitors, prostaglandins or mucosal protective agents prior to study in 2 weeks
* Patient who cannot interrupt steroid, non-steroid anti-inflammatory drugs or aspirin during treatment
* Allergic or hypersensitive to any of the ingredients in the test products
* Pregnant or lactating female
* Patients who have abnormal baseline laboratory test result
* Patients taking other investigational drugs within 30 days prior to the study.
* Patients with Zollinger-Ellison syndrome
* Patients that investigators consider ineligible for this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
A percentage of subjects showed moderate improvement of stomach erosions by the endoscopy | 2 weeks
  The definition of "moderate improvement" is the subjects showed score changed from 2-4 to 1 or from 4 to 2.
  [score 1(normal) : no erosion, score 2(mild) : 1-2 erosions, score 3(moderate) : 3-5 erosions, score 4(severe) : 6 or more erosions]

SECONDARY OUTCOMES:
A percentage of subjects showed significant improvement of stomach erosions by the endoscopy | 2 weeks
  The definition of "significant improvement" is the subject showed score changed from 2-4 to 1.
  [score 1(normal) : no erosion, score 2(mild) : 1-2 erosions, score 3(moderate) : 3-5 erosions, score 4(severe) : 6 or more erosions]
A percentage of subjects showed improvement of edema rating scale | 2 weeks
  The definition of "improvement" is the subjects showed score changed from 2 to 1.
A percentage of subjects showed improvement of erythema rating scale | 2 weeks
  The definition of "improvement" is the subjects showed reduction ratio of score changed 50% or more.
A percentage of subjects showed improvement of hemorrhage rating scale | 2 weeks
  The definition of "improvement" is the subjects showed reduction ratio of score changed 50% or more.
A percentage of subjects showed improvement of gastric symptom rating scale | 2 weeks
  The definition of "improvement" is the subjects showed reduction ratio of score changed 50% or more.
Adverse Events | 2 weeks
Lab results(Hematology, Blood chemistry, Urinalysis) | 2 weeks
The results of physical examinations and Vital signs(body temperature, pulse) | 2 weeks
EKG results | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hyo Jin Park, MD, Ph.D, Principal Investigator — Yonsei University, Gangnam Severance Hospital of Korea
Locations (14):
- South Korea (14):
  - Inje University, Busan Paik Hospital of Korea, Busan
  - Keimyung University, Dongsan Medical Center of Korea, Daegu
  - Wonkwang University, Hospital of Korea, Iksan-si
  - Seoul National University, Bundang Hospital of Korea, Seongnam-si
  - Chungang University, Hospital of Korea, Seoul
  - Ewha Womans University, Medical Center of Korea, Seoul
  - Inje University, Seoul Paik Hospital of Korea, Seoul
  - Kankbuk Samsung Medical Center of Korea, Seoul
  - Korea University, Guro Hospital of Korea, Seoul
  - Seoul National University, Hospital of Korea, Seoul
  - Soonchunhyang University, Seoul Hospital of Korea, Seoul
  - The Catholic University, Seoul St. Mary's Hospital of Korea, Seoul
  - Yonsei University, Gangnam Severance Hospital of Korea, Seoul
  - Ajou University, Medical Center of Korea, Suwon